CLINICAL TRIAL: NCT06323993
Title: The Clinical Outcomes of Lateral Sinus Floor Elevation With Different Window Preparation Approaches: a Retrospective Study
Brief Title: The Effect of Different Window-preparation Approaches on the Clinical Outcomes of Lateral Sinus Floor Elevation
Status: Completed | Type: Observational
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Guoli Yang, Director of Implantology Department, The Dental Hospital of Zhejiang University School of Medicine
Other Study IDs: 2021-115
Record Dates: First submitted 2023-09-03; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Dental Implantation; Cone-Beam Computed Tomography; Surgical Procedure, Unspecified; Maxillary Sinus Floor Augmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Piezoelectric osteotomy: This group used piezoelectric osteotomy (exposure) to prepare the lateral window acceding maxillary sinus
  Interventions: Procedure: Piezoelectric osteotomy
- Round Bur: This group used round bur (control) to prepare the lateral window acceding maxillary sinus

INTERVENTIONS:
Procedure: Piezoelectric osteotomy — The piezoelectric technique, another window preparation procedure that does not use a round bur, was first introduced to LSFE in 2001 for its high accuracy of osteotomy and low rate of membrane perforation. Later studies demonstrated that the operation time, postoperative reactions, and perforation rate of this procedure are considered to be acceptable compared with rotary bur. Moreover, the piezoelectric technique allows for the lateral bone window to be cut and preserved relatively completely.
  Groups: Piezoelectric osteotomy

SUMMARY:
This study retrospectively evaluated the effect of two different lateral window preparation techniques on peri-implant bone augmentation for patients who underwent lateral sinus floor elevation with simultaneous implant placement using two-dimensional and three-dimensional radiographic results, with special emphasis placed on the stability of the graft material after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* one or more maxillary posterior teeth were missing, and the healing time was more than 3 months;
* complete basic information and detailed operation records;
* available CBCT images before surgery, immediately after surgery, and 6 months after surgery;
* RBH ≤6 mm shown by CBCT at T0 at the site of the missing tooth；
* no systematic diseases and no untreated periapical disease or periodontal disease before surgery.

Exclusion Criteria:

* (1) maxillary lesions have not been properly treated；
* present or past medication of bisphosphonates;
* pregnancy or lactation;
* present or past radiotherapy of head and neck cancer within 5 years;
* acute and chronic inflammation in the maxillary sinus;
* in need of additional vertical or horizontal bone augmentation besides LSFE with endo-sinus graft materials;
* heavy smoker (>20 cigarettes/day at the time of surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects were selected among patients who have received LSFE with graft materials with simultaneous implant placement from November 2018 to June 2021 in the Department of Implantology at the Affiliated Hospital of Stomatology, Zhejiang University School of Medicine, China.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Apical bone height | Immediately after surgery, and 6 months after surgery
  The distance (mm) from the implant apex to the most apical position of the graft material along the longitudinal axis of the implant
Endo-sinus bone gain | Immediately after surgery, and 6 months after surgery
  The distance (mm) from the level of the sinus floor (middle of the buccal level and palatal level) to the level of the most apical position of the graft material along the longitudinal axis of the implant
Palatal bone height | Immediately after surgery, and 6 months after surgery
  The vertical distance (mm) from the api- cal margin of the implant shoulder on the palatal side straight up to the position of the most apical position of the graft material
Buccal bone height | Immediately after surgery, and 6 months after surgery
  The vertical distance (mm) from the api- cal margin of the implant shoulder on the buccal side straight up to the position of the most apical position of the graft material
Augmentation volume | Immediately after surgery, and 6 months after surgery
  The volume of the endo-sinus reconstructed graft materials

SECONDARY OUTCOMES:
Perforation incidence | During the surgery
  Sinus perforation was determined by direct visualization and the Valsalva maneuver during the surgery process.
Early implant loss | 6 months after surgery
  Early implant loss was defined as an implant show- ing clinical mobility prior to the placement of the abutment
Lateral window length | Immediately after surgery, and 6 months after surgery
  the distance between the edges of lateral window caused by the lateral antrostomy
Lateral bone length | Immediately after surgery, and 6 months after surgery
  the length of the bone window ob- tained by piezoelectric osteotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Stomatology Hospital, School of Stomatology, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China